CLINICAL TRIAL: NCT05722496
Title: Interval Versus Continous Intradialytic Training on Muscla Quality Index and Functional Capacity in Hemodialysis Patients
Brief Title: Difference Between Interval and Continous Intradialytic Exercise on Functional Capacity in Hemodialysis Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Saber Mansour El-Sayed, assistant lecturer at department of cardiovascular, respiratory and geriatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111118
Record Dates: First submitted 2023-01-23; First posted 2023-02-10 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hemodialysis Complication

STUDY DESIGN:
Intervention Model Description: Patients will be assigned randomly by computerized block randomization into two groups:Group (A): 30 patients aged between 45 - 55 years old will participate in 8 weeks of aerobic exercise in the form of high intensity interval training (HIIT) intradialytic pedaling exercise plus hemodialysis (3 sessions per week).
  Group (B): 30 patients aged between 45- 55 years old will participate in 8 weeks of aerobic exercise in the form of moderate intensity continous training (MICT) intradialytic pedaling exercise plus hemodialysis (3 sessions per week).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: block randomization and envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training Group (Group A) (Experimental): Each training session consist of three parts of 30 minutes:
  * Warm up (5 minutes) free active exercise of the lower extremities,
  * Training continued with three exercise intervals lasting 3 min each, at an exercise intensity of 85%-95% of HRpeak equalling 15-17 on the Borg scale. Each interval was separated by 4 min of active breaks at an intensity of 60%-70% of HRpeak.
  * Cool down (5 minutes) free exercise of lower extremities. Training program will last for 8 weeks with frequency 3times / week.
  Interventions: Other: Aerobic pedaling exercise
- Moderate intensity continous training group (Group B) (Experimental): Each training session consist of three parts of 30 minutes:
  * Warm up (5 minutes) free active exercise of the lower extremities,
  * Training continued with cycling at low-to-moderate exercise intensity of 50%-60% of HRpeak, representing 11-13 on the Borg scale.
  * Cool down (5 minutes) free exercise of lower extremities. Training program will last for 8 weeks with frequency 3times / week.
  Interventions: Other: Aerobic pedaling exercise

INTERVENTIONS:
Other: Aerobic pedaling exercise — aerobic exercise in the form of leg pedaling exercise in semi-supine position using leg ergometer by different intensities

SUMMARY:
The goal of this study is to find out the effect of interval versus continous intradialytic training on muscle quality index and functional capacity in Hemodialysis patients. The main question it aims to answer is:

Does interval versus continous intradialytic training have an effect on muscle quality index and functional capacity in hemodialysis patients? Patients will be assigned randomly by computerized block randomization into two groups:Group (A): 30 patients will participate in 8 weeks of aerobic exercise in the form of high intensity interval training (HIIT) intradialytic pedaling exercise plus hemodialysis (3 sessions per week).Group (B): 30 patients will participate in 8 weeks of aerobic exercise in the form of moderate intensity continous training (MICT) intradialytic pedaling exercise plus hemodialysis (3 sessions per week) . primary and secondary variables will be measured before starting treatment and after completion (after 2 months )

DETAILED DESCRIPTION:
Individuals with CKD (both predialysis and ESRD) may be at greater risk of sarcopenia given the combined reductions in physical function, skeletal muscle performance and skeletal muscle mass.

Study include sixty male patients on hemodialysis for 1-3 years aged from 45 to 55 years old selected from hemodialysis unit at National Institute of Urology and Nephrology. Before starting treatment , patients will fill consent form and the study aims and procedure will be explained to each patient . study include Sixty male patients on hemodialysis for 1-3 years aged from 45 to 55 years old selected from hemodialysis unit at National Institute of Urology and Nephrology. Patients will be assigned randomly by computerized block randomization into two groups:Group (A): 30 patients will participate in 8 weeks of aerobic exercise in the form of high intensity interval training (HIIT) intradialytic pedaling exercise plus hemodialysis (3 sessions per week).Group (B): 30 patients will participate in 8 weeks of aerobic exercise in the form of moderate intensity continous training (MICT) intradialytic pedaling exercise plus hemodialysis (3 sessions per week) Karvonen formula will be used to calculate training heart rate THR= RHR+ (HRmax - RHR) 65%-80% AS HRmax = 220-Age patients of HIIT will perform aerobic exercise in the form of leg pedaling exercise in semi-supine position using leg ergometer at high intensity 85%-95% of HRpeak with 4 min of active breaks at an intensity of 60%-70% of HRpeak. . Exercise will be done at the first 2 hours of dialysis (to avoid dialysis hypotension episodes).

patients of MICT will perform aerobic exercise in the form of leg pedaling exercise in semi-supine position using leg ergometer at moderate intensity 50%-60% of HRpeak . Exercise will be done at the first 2 hours of dialysis (to avoid dialysis hypotension episodes).

primary and secondary variables will be measured before starting treatment and after completion (after 2 months )

ELIGIBILITY:
Inclusion Criteria:

1. Age between 45- 55 years.
2. Male sex included.
3. Patients with grade 5 chronic renal failure on hemodialysis.
4. Patients are on hemodialysis for 1-3 years.
5. Body mass index (BMI) range from 25-34.9 Kg/m2.
6. They will be medically and psychologically stable.
7. Receiving their physician-prescribed pharmacotherapy regularly.
8. Agree to participate by signing an informed consent form.

Exclusion Criteria:

1. Inability to comprehend and follow instructions as in dementia or speech problems such as dysphasia.
2. Patients with unstable angina, uncontrolled cardiac arrhythmia, decompensated heart failure, persistent systolic blood pressure (BP) greater than 200 mmHg, persistent diastolic BP greater than 120 mmHg, acute pericarditis or myocarditis.
3. Acute systemic infection.
4. Presence of malignant disease.
5. Patients with Diabetes Mellitus.
6. Patients with Lupus Nephritis.
7. Patients with chronic obstructive lung disease, restrictive lung disease or chronic chest infection.
8. Severe obesity (BMI > 35).
9. Chronic inflammatory orthopedic disorders and rheumatoid arthritis.
10. Patients with muscle injuries or neuromuscular disorders (muscular dystrophy, myasthenia gravis, myopathy, multiple sclerosis and peripheral neuropathy).

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
muscle quality index | 2 months
  The MQI was quantified using a timed sit-to-stand test, body mass, and leg length to calculate a power index that is expressed in watts (W). The MQI was calculated as follows:
  QI (Watts) = ((Leg length×0.4) ×Bodymass×gravity×10) ∕ Time taken for (sit to stand 5 times) Body mass will be measured using a digital scale. Leg length will be taken using tape measure to measure the distance (in meters) from the greater trochanter of the femur to the lateral malleolus, measured from standing position . BY using a stopwatch, sit-to-stand time will be calculated as the time to stand from a seated position and return to sitting consecutively five times. The use of arms not allowed during the sit-to-stand test. Acceleration of gravity (9.8 m/s2).
  After measuring leg length, body mass and time for sit to stand, all these data will be written in the previous equation to calculate muscle quality index and expressed in watts (W).
six minute walk test | 2 months
  Six minute walk test (6MWT) to assess physical functional capacity (using stopwatch, colored tape to mark starting line and end line of corridor) Using a stopwatch, assess physical functional capability. The 6MWT will be conducted indoors along a 30 m long, level, straight, enclosed hallway, with the length of the corridor indicated with brightly coloured tape at the beginning and end lines. Subjects will be advised to walk as far as possible from end to end of the corridor without jogging or running, and to cover as much distance as feasible in the 6 minute time limit . This test was performed at the beginning of treatment and at the end of treatment program (8 weeks) to assess functional performance difference.

CONTACTS AND LOCATIONS:
Overall Officials: hala m ezz eldeen, professor, Study Director — department of cardiovascular, respiratory and geriatrics disorders
Locations (1):
- Faculty of physical therapy, cairo university, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No
after completion of the study and publication, data will be available for other researchers